CLINICAL TRIAL: NCT06100107
Title: Mirror Visual Feedback as Therapeutic Modality in Unilateral Upper Extremity Complex Regional Pain Syndrome Type I
Brief Title: Mirror Therapy in Complex Regional Pain Syndrome Type I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Rudolf Cerny, Senior Investigator, University Hospital, Motol
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EK-1288/14
Record Dates: First submitted 2023-10-12; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Complex Regional Pain Syndrome Type I
MeSH Terms: conditions — Complex Regional Pain Syndromes

STUDY DESIGN:
Intervention Model Description: Specifically, the study employs a half cross-over design. Group A begins with the intervention, while Group B starts with a control period of equal length, followed by the intervention. This design facilitates comparisons both between the groups and within Group B across the two periods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Mirror Therapy (Experimental): Group A carried out a ten-minute Mirror Therapy exercise daily, for a total duration of six weeks.
  Interventions: Other: Mirror Therapy exercise
- Group B - control period followed by Mirror Therapy (Experimental): Group B acted as a control group for six weeks (no Mirror Therapy) followed by six weeks of Mirror Therapy with the same characteristics as Group A.
  Interventions: Other: Mirror Therapy exercise

INTERVENTIONS:
Other: Mirror Therapy exercise — Mirror Therapy for the upper limb involves the use of a mirror to create a reflected image of the unaffected arm, making it appear as if both arms are moving symmetrically. During the therapy, the patient places their affected arm behind the mirror and their unaffected arm in front. While focusing on the mirror reflection, the patient performs various movements with the unaffected arm, giving the illusion that the affected arm is moving normally.
  Other Names: Mirror visual feedback exercise

SUMMARY:
The aim is to evaluate the efficacy of Mirror Therapy on pain reduction and hand function in subjects with unilateral upper extremity Complex Regional Pain Syndrome Type I.

DETAILED DESCRIPTION:
Subjects were randomly divided into two groups. Group A carried out a ten-minute Mirror Therapy exercise daily, for a total duration of six weeks. Group B acted as a control group for six weeks followed by six weeks of Mirror Therapy with the same characteristics as Group A. Upper extremity active range of motion, strength, dexterity, limb volume, right-left temperature difference, and health-related quality of life were evaluated before and after each period. Daily records on the visual analogue scale were used for pain evaluation. Effectiveness was calculated using mixed-effects modelling for between-group comparisons and within-group variability and identifying significant predictors.

ELIGIBILITY:
Inclusion Criteria:

- diagnosis of CRPS I based on the Budapest criteria

Exclusion Criteria:

* failure to meet the diagnostic Budapest clinical criteria for CRPS I
* previous use of Mirror Therapy prior to the commencement of this study
* substantial difficulties in cooperation
* a significant change to the subjects' treatment regimen, outside of the study design

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-09-09 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2016-01-15 (Actual)

PRIMARY OUTCOMES:
Pain perception | Recordings performed every day from day 0 to day 42 (Group A) and from day 0 to day 84 (Group B); Follow-up on day 72 (Group A) and day 114 (Group B).
  The participants in both groups made daily accounts of their pain level using 10 cm long visual analog scale (VAS) at rest as well as typical pain level during hand movement.
Active Range of Motion | On day 0 (Group A, Group B); on day 42 (Group A, Group B); on day 84 (Group B)
  Three attributes were measured: maximal active range of wrist flexion and extension (°) determined with goniometer measuring the angle between forearm and metacarpal bones
Strength | On day 0 (Group A, Group B); on day 42 (Group A, Group B); on day 84 (Group B)
  The outcome parameter is the highest pressure (bar) performed during one maximal grip.
Dexterity | On day 0 (Group A, Group B); on day 42 (Group A, Group B); on day 84 (Group B)
  Dexterity was evaluated by using a nine-hole PegBoard. The time taken to complete this task was measured.
Volume of hand and forearm | On day 0 (Group A, Group B); on day 42 (Group A, Group B); on day 84 (Group B)
  The volumetric measurements are based on the principle of water displacement.
Temperature | On day 0 (Group A, Group B); on day 42 (Group A, Group B); on day 84 (Group B)
  Temperature was measured bilaterally in the thenar area using an infrared thermometer.
Health-related Quality of Life | On day 0 (Group A, Group B); on day 42 (Group A, Group B); on day 84 (Group B)
  Determined using the European Quality of Life-5 Dimensions-3 Levels questionnaire. A range of 0-100% is used, where a higher score means a better outcome.